CLINICAL TRIAL: NCT02957604
Title: Evolocumab Pregnancy Exposure Registry: An OTIS Pregnancy Surveillance Study
Brief Title: Evolocumab Pregnancy Exposure Registry
Status: Terminated | Type: Observational
Sponsor: Amgen (Industry)
Collaborators: Organization of Teratology Information Specialists (OTIS) Research Center - tel: 1-866-626-6847 or www.mothertobaby.org (Unknown)
Responsible Party: Sponsor
Other Study IDs: 20150338
Record Dates: First submitted 2016-10-26; First posted 2016-11-08 (Estimated); Last update posted 2020-12-17 (Actual); Status verified 2020-12

CONDITIONS: Hypercholesterolemia; ASCVD; Pregnancy
Keywords: Pregnancy; Cardiovascular Diseases; High serum cholesterol; FH; ASCVD
MeSH Terms: conditions — Hypercholesterolemia; Cardiovascular Diseases | interventions — evolocumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Specific Evolocumab-Exposed Cohort: Women diagnosed with Atherosclerotic Cardiovascular Disease (ASCVD), or hypercholesterolemia associated with Familial Hypercholesterolemia (FH), who were exposed to Evolocumab (Repatha) during pregnancy
  Interventions: Drug: evolocumab
- Comparison Group I: Women diagnosed with Atherosclerotic Cardiovascular Disease (ASCVD), or hypercholesterolemia associated with Familial Hypercholesterolemia (FH) who were not exposed to Evolocumab during pregnancy
- Comparison Group II: A general comparison group of pregnant women who have not been diagnosed with Atherosclerotic Cardiovascular Disease (ASCVD), or hypercholesterolemia associated with Familial Hypercholesterolemia (FH), and who were not exposed to Evolocumab during pregnancy.
- General Evolocumab-Exposed Case Series: Women who were exposed to Evolocumab (Repatha) but do not fulfill eligibility criteria for the Specific Evolocumab-Exposed Cohort
  Interventions: Drug: evolocumab

INTERVENTIONS:
Drug: evolocumab — Pregnant women exposed to evolocumab. Evolocumab is not administered in this non-interventional study.
  Other Names: Repatha
  Groups: General Evolocumab-Exposed Case Series; Specific Evolocumab-Exposed Cohort

SUMMARY:
This is a prospective observational registry study to evaluate fetal, infant and childhood outcomes in women exposed to evolocumab during pregnancy

DETAILED DESCRIPTION:
This pregnancy registry will be conducted by University of California Research Center for the Organization of Teratology Information Specialists (OTIS) which is a network of university and health department based telephone information centers serving pregnant women and healthcare providers throughout North America. Participants will be enrolled on an ongoing basis through year 10 of the study and each will be followed from the time they enroll, through the 5-year postnatal follow up period for an overall study period of 15 years. Participants are recruited concurrently from callers to OTIS centers, from healthcare providers and through direct to consumer marketing efforts.

ELIGIBILITY:
Inclusion Criteria:

* For all groups: Qualified subjects will agree to the conditions and requirements of the study including the interview schedule, release of medical records, the physical examination of live born infants, and 5 years of follow-up.
* For the Specific Evolocumab-Exposed Cohort: Currently pregnant women (maternal report validated by medical records) diagnosed with ASCVD, or hypercholesterolemia associated with FH who have been exposed to evolocumab for any number of days, at any dose, and at any time from the first day of the LMP up to and including the end of pregnancy.
* For Comparison Group I: Currently pregnant women (maternal report validated by medical records) diagnosed with ASCVD, or hypercholesterolemia associated with FH but who were not exposed to evolocumab during pregnancy or any time within 90 days prior to the first day of the LMP.
* For Comparison Group II: Currently pregnant women not diagnosed with ASCVD, or hypercholesterolemia associated with FH who have not been exposed to evolocumab during pregnancy or any time within 90 days prior to the first day of the LMP, and who have no exposure to any known human teratogens as determined by the OTIS Research Center
* For General Evolocumab-Exposed Case Series group: Women with exposure to evolocumab during pregnancy who do not meet the criteria for the Specific Evolocumab-Exposed cohort for reasons including (but not limited to): they do not have ASCVD and/or hypercholesterolemia associated with FH (off-label use), they were exposed to evolocumab but the pregnancy has already completed, they enrolled in the cohort study with a previous pregnancy, or they already have a prenatal diagnosis of a major birth defect

Exclusion Criteria:

For all groups except the General Evolocumab Exposed Case Series Group:

* Women who first contact the Registry after prenatal diagnosis of a major structural defect
* Women who were exposed to a different PCSK9 inhibitor during their current pregnancy or at any time within 5 half-lives prior to the first day of the LMP
* Women who have enrolled in this Registry with a previous pregnancy

Ages: 1 Year to 100 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Pregnant women diagnosed with ASCVD or hypercholesterolemia associated with FH and pregnant women who have been exposed to Evolocumab (Repatha) during pregnancy and who reside in the U.S. or Canada
Sampling Method: Non-Probability Sample
Enrollment: 140 (Actual)
Dates: Start 2016-12-22 (Actual); Primary Completion 2020-09-02 (Actual); Study Completion 2020-09-02 (Actual)

PRIMARY OUTCOMES:
Rate of major structural defects | Up to 1 year of age
  Rate of major structural defects, defined and classified by the Centers for Disease Control and Prevention (CDC) Metropolitan Atlanta Congenital Defects Program (MACDP) 6 Digit Code Defects List coding manual (CDC, 2007)

SECONDARY OUTCOMES:
Pregnancy Outcome: Rate of spontaneous abortion | Up to 19 wks post LMP
  Rate of spontaneous abortion where spontaneous abortion is defined as non-deliberate fetal death which occurs prior to 19 completed weeks post-last menstrual period (LMP)
Pregnancy Outcome: Rate of elective abortion | Through 9 month pregnancy period
  Rate of elective abortion where elective abortion is defined as deliberate termination of pregnancy at any time in gestation
Pregnancy Outcome: Rate of stillbirth | At or after 19 completed weeks post LMP
  Rate of stillbirth where stillbirth is defined as non-deliberate fetal death anytime in gestation at or after 19 completed weeks post-LMP
Pregnancy Outcome: Rate of premature delivery | Prior to 37 weeks of gestation
  Rate of premature delivery where premature delivery is defined as live birth prior to 37.0 weeks gestation as counted from LMP (or ultrasound adjusted date)
Infant Outcome: Rate of minor structural defects | Between birth and 12 months post natal
  Rate of minor structural defects where a minor structural defect is defined as a structural anomaly which has neither cosmetic nor functional significance to the child.
Infant Outcome: Rate of small for gestational age | At birth
  Rate of small for gestational age where small for gestational age is defined as birth size (weight, length, or head circumference) less than/equal to the 10th centile for sex and gestational age using standard pediatric CDC growth curves for full term or preterm infants
Infant Outcome: Rate of postnatal growth deficiency | Up to 1 year of age
  Rate of postnatal growth deficiency where postnatal growth deficiency is defined as postnatal size (weight, length, or head circumference) less than/equal to the 10th centile for sex and age using standard pediatric growth curves, and adjusted for postnatal age for premature infants if the postnatal measurement is obtained at less than 1 year of age.
Infant Outcome: Rate of postnatal hospitalizations | Through 5 years postnatal
  Rate of postnatal hospitalizations as assessed throughout the 5-year postnatal follow-up period.
Infant Outcome: Rate of infant reactions to scheduled vaccinations | Through 5 years postnatal
  Rate of infant reactions to scheduled vaccinations as assessed throughout the 5-year postnatal follow-up period.
Infant Outcome: Infant response to IgG-tetanus antibody | Between 6-12 months of age
  Infant response to IgG-tetanus antibody as a biological marker to evaluate humoral immune response via a standardized assay test.
Infant Outcome: Adverse neurodevelopment outcomes | Between 16 months to 17 months 30 days of age and between 3.5-5 years of age
  Adverse neurodevelopmental outcomes as assessed during 2 periods (between 16 months to 17 months 30 days of age and between 3.5-5 years of age) via standardized tests of performance
Breastfeeding/Lactation Outcome: Proportion of women who breastfed | Through 6 weeks post delivery
  Proportion of women who breastfed (at all) in the first 6 weeks after delivery
Breastfeeding/Lactation Outcome: Proportion who breastfed exclusively | Through the first 2 weeks postnatal
  Among women who breastfed (in the first 6 weeks after delivery), the proportion who breastfed exclusively during the first 2 weeks of life
Infant Outcome: Pattern of minor structural defects | Between birth and 12 months postnatal
  Pattern of minor structural defects where a minor structural defect is defined as a structural anomaly which has neither cosmetic nor functional significance to the child and a pattern is defined as the same 3 or more minor structural defects in 2 or more children.
Infant Outcome: Rate of postnatal serious infections | Through 5 years postnatal
  Rate of postnatal serious infections as assessed throughout the 5-year postnatal follow-up period.

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data sharing requests relating to this study will be considered beginning 18 months after the study has ended and either 1) the product and indication (or other new use) have been granted marketing authorization in both the US and Europe or 2) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this study.
Access Criteria: Qualified researchers may submit a request containing the research objectives, the Amgen product(s) and Amgen study/studies in scope, endpoints/outcomes of interest, statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). In general, Amgen does not grant external requests for individual patient data for the purpose of re-evaluating safety and efficacy issues already addressed in the product labelling. Requests are reviewed by a committee of internal advisors, and if not approved, may be further arbitrated by a Data Sharing Independent Review Panel. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement. This may include anonymized individual patient data and/or available supporting documents, containing fragments of analysis code where provided in analysis specifications. Further details are available at the link below.
URL: https://www.amgen.com/datasharing

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com